CLINICAL TRIAL: NCT04209270
Title: Breathing Pattern, Work of Breathing and Gas Exchange in Patients With Acute Respiratory Distress Syndrome During the Spontaneous Breathing Trial
Brief Title: Breathing Pattern, WOB and Gas Exchange in Patients With Acute Respiratory Distress Syndrome During the Spontaneous Breathing Trial
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sanatorio de la Trinidad Mitre (Other)
Responsible Party: Principal Investigator, María Lucía Gimenez, RT, Sanatorio de la Trinidad Mitre, Sanatorio de la Trinidad Mitre
Other Study IDs: WOB in ARDS
Record Dates: First submitted 2019-12-19; First posted 2019-12-24 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Work of Breathing; ARDS; Weaning Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is little evidence about the mechanical characteristics and muscular function in patients with Acute Respiratory Distress Syndrome (ARDS) at the time of weaning of the mechanical ventilation, as well as the behavior of the mechanical properties, breathing pattern, muscular effort, and gas exchange during a successful and failed spontaneous breathing trial.

DETAILED DESCRIPTION:
The study of the respiratory system (RS) mechanics in patients with ARDS has been focused on the initial phase of ventilatory support, with few studies observing the weaning in mechanical ventilation.The RS in patients with ARDS is characterized by a greater or lesser degree of low functional residual capacity (FRC) in relation to normal.

At the time of performing a spontaneous breathing trial, these mechanical characteristics determine the need to develop a high transpulmonary pressure during each breath, with high work of breathing (WOB) to achieve adequate alveolar ventilation.

Inspiratory muscle weakness could alter the ability to generate the necessary transpulmonary pressure over time according to the loads imposed at the time of performing a spontaneous breathing trial, with the consequent development of fatigue and ventilatory failure.

This is why the investigators propose to evaluate the association between elastic WOB and the failure of the spontaneous breathing trial.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* requiring mechanical ventilation for more than 12 hours
* moderate/ severe ARDS according to Berlin Definition
* able to make a Spontaneous Breathing Trial according to the institution protocol

Exclusion Criteria:

* pregnant patients
* history of neuromuscular disease
* patients in palliative care
* bronchopleural fistula
* contraindication of measurement of esophageal pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will meassure adult, ARDS, Intensive Care Unit patients that are able to perform a Spontaneous Breathing Trial.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Spontaneous breathing Trial | During 60 minutes after inclusion or until the patient fails to breathe spontaneously
  Period of time in which the patient breathes spontaneously

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Fredes, RT, Principal Investigator — Sanatorio de la Trinidad Mitre
Locations (1):
- Sanatorio de la Trinidad Mitre, Buenos Aires, Argentina